CLINICAL TRIAL: NCT02625051
Title: Randomized Controlled Clinical Trial Comparing Ureteroscopic to Percutaneous Removal for the 1-2 cm Calculus Measuring Quality of Life as the Primary Outcome
Brief Title: Quality of Life in Kidney Stone Patients Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHR15-17595; P20DK100863 (NIH)
Record Dates: First submitted 2015-12-04; First posted 2015-12-09 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Kidney Calculi; Quality of Life
MeSH Terms: conditions — Kidney Calculi | interventions — Ureteroscopy; Nephrolithotomy, Percutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ureteroscopy (Active Comparator): Kidney stone of participants in this arm will be treated with ureteroscopy (URS). A ureteral stent will be inserted at the end of the procedure.
  Interventions: Procedure: Ureteroscopy
- Percutaneous nephrolithotomy (Active Comparator): Kidney stone of participants in this arm will be treated with percutaneous nephrolithotomy (PNL). A percutaneous nephrostomy tube will be inserted at the end of the procedure.
  Interventions: Procedure: Percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: Ureteroscopy — Under general anesthesia, the patient is placed in the lithotomy position. All procedures are performed under direct videoscopic and fluoroscopic guidance. Fluoroscopic screening is utilized using a mobile multidirectional C-arm fluoroscopy unit. A safety guide-wire is then placed into renal pelvis, followed by a ureteral access sheath to maintain low intra-renal pressure, and to facilitate the procedures. Using flexible ureteroscope, renal or proximal ureteral stone is identified and fragmented with a holmium laser. Basket extraction of residual fragments is done until visual complete clearance of stone fragments is achieved.
  Other Names: URS
  Arms: Ureteroscopy
Procedure: Percutaneous nephrolithotomy — Under general anesthesia, an open-ended 5 french ureteral exchange catheter is placed into the ipsilateral ureter under cystoscopic guidance. The patient is then safely turned and secured in the prone position. Percutaneous renal access is obtained under ultrasonographic or fluoroscopic guidance. Either a 24 or 30 french sheath is advanced in the kidney and nephroscopy is performed with a rigid offset nephroscope. Stone fragmentation is accomplished using a dual CyberWand lithotripter or holmium laser lithotripsy. Flexible nephroscopy is performed to look for possible residual fragments and basket extraction is done for complete clearance of stone.
  Other Names: PNL
  Arms: Percutaneous nephrolithotomy

SUMMARY:
This is a prospective randomized study, comparing quality of life in renal stone patients undergoing surgical treatment with ureteroscopy (URS) versus percutaneous nephrolithotomy (PNL).

DETAILED DESCRIPTION:
In United States, the prevalence of renal stone is 8.8% with slight predomination in male than female. They can be symptomatic marked by symptoms of flank pain, hematuria or urinary tract infection, or completely asymptomatic and incidentally discovered. Three modalities are accepted as treatment options for renal stone, including shockwave lithotripsy (SWL), percutaneous nephrolithotomy (PNL) and ureteroscopy (URS). While some standard guidelines were proposed for appropriate treatment selection with regard to stone size, no recommendations or guidelines exist for the surgical management of 1-2 cm renal stones. Both PNL and URS are equally accepted as treatment options for stones at this size. The selection of either procedure currently is left to the treating surgeon can be influenced by anatomical or stone factors as well as patient preference. For URS, frequent requirement for postoperative ureteral stents may result in significant morbidity and a detriment to quality of life owing to irritating bladder symptoms caused by the stent itself. PNL rarely requires postoperative ureteral stent but it may bring longer operative time and hospitalization. PNL therefore may be a treatment option that preserves quality of life compared to URS for patients presenting with the 1-2 cm sized kidney or ureteral stone.

One reasonable way to evaluate efficacy of treatment options is to assess patient's quality of life resultant from the selected modality. Quality of life for renal stone formers is an important but under-studied facet of nephrolithiasis management that should be incorporated into clinical decision making.

The short form-36 health survey questionnaire (SF-36) is a patient-reported survey of health status. It has been validated and is commonly used to determine the efficacy of a given health treatment in many settings, including urologic intervention. The Ureteral Stent Symptom Questionnaire (USSQ) is a validated and widely accepted instrument to evaluate the impact of ureteral stents on quality of life. The investigators plan to use these two questionnaires as a standard outcome measurement to compare impact on quality of life in patients randomized to undergo two different modalities (PNL versus URS) of stone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a renal or proximal ureteral stone measuring 1-2 cm in size on preoperative ultrasound, computed tomography, or plain radiographic imaging

Exclusion Criteria:

* Serious illness likely to cause death within the next 5 years, so as to exclude significant metabolic derangements that might lead to adverse surgical outcome.
* Stones with measured size larger than 2 cm or smaller than 1 cm.
* Patients with ureteral or renal anatomy or stones located in a position judged to be unsafe for randomization.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change of overall quality of life (QOL) score as measured by Short form-36 (SF-36) Questionnaire at early postoperative period | Change from baseline score at 1 week after surgery
  This instrument consisted of 36 questions with response ranging from 0 (poor QOL) to 100 (best QOL).

SECONDARY OUTCOMES:
Change of overall quality of life (QOL) score as measured by Ureteral Stent Symptom Questionnaire (USSQ) at early postoperative period | Change from baseline score at 1 week after surgery
  This instrument consisted of 38 questions in 6 non-uniformed categories with response ranging from the least (best QOL) to the most (poor QOL).

OTHER OUTCOMES:
Change of overall quality of life (QOL) score as measured by Short form-36 (SF-36) Questionnaire at late postoperative period | Change from baseline score at 3 months after surgery
  This instrument consisted of 36 questions with response ranging from 0 (poor QOL) to 100 (best QOL).
Change of overall quality of life (QOL) score as measured by Ureteral Stent Symptom Questionnaire (USSQ) at late postoperative period | Change from baseline score at 3 months after surgery
  This instrument consisted of 38 questions in 6 non-uniformed categories with response ranging from the least (best QOL) to the most (poor QOL).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chi, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Scales CD Jr, Smith AC, Hanley JM, Saigal CS; Urologic Diseases in America Project. Prevalence of kidney stones in the United States. Eur Urol. 2012 Jul;62(1):160-5. doi: 10.1016/j.eururo.2012.03.052. Epub 2012 Mar 31. PMID 22498635
- [Background] Pearle MS, Calhoun EA, Curhan GC; Urologic Diseases of America Project. Urologic diseases in America project: urolithiasis. J Urol. 2005 Mar;173(3):848-57. doi: 10.1097/01.ju.0000152082.14384.d7. PMID 15711292
- [Background] Tiselius HG, Ackermann D, Alken P, Buck C, Conort P, Gallucci M; Working Party on Lithiasis, European Association of Urology. Guidelines on urolithiasis. Eur Urol. 2001 Oct;40(4):362-71. doi: 10.1159/000049803. PMID 11713390
- [Background] Kumar A, Kumar N, Vasudeva P, Kumar Jha S, Kumar R, Singh H. A prospective, randomized comparison of shock wave lithotripsy, retrograde intrarenal surgery and miniperc for treatment of 1 to 2 cm radiolucent lower calyceal renal calculi: a single center experience. J Urol. 2015 Jan;193(1):160-4. doi: 10.1016/j.juro.2014.07.088. Epub 2014 Jul 24. PMID 25066869
- [Background] Duvdevani M, Chew BH, Denstedt JD. Minimizing symptoms in patients with ureteric stents. Curr Opin Urol. 2006 Mar;16(2):77-82. doi: 10.1097/01.mou.0000193375.29942.0f. PMID 16479208
- [Background] Haleblian G, Kijvikai K, de la Rosette J, Preminger G. Ureteral stenting and urinary stone management: a systematic review. J Urol. 2008 Feb;179(2):424-30. doi: 10.1016/j.juro.2007.09.026. PMID 18076928
- [Background] Kirac M, Bozkurt OF, Tunc L, Guneri C, Unsal A, Biri H. Comparison of retrograde intrarenal surgery and mini-percutaneous nephrolithotomy in management of lower-pole renal stones with a diameter of smaller than 15 mm. Urolithiasis. 2013 Jun;41(3):241-6. doi: 10.1007/s00240-013-0552-0. Epub 2013 Mar 13. PMID 23483226
- [Background] Perez-Fentes DA, Gude F, Blanco B, Freire CG. Percutaneous nephrolithotomy: short- and long-term effects on health-related quality of life. J Endourol. 2015 Jan;29(1):13-7. doi: 10.1089/end.2014.0081. PMID 24708396
- [Background] Barnes KT, Bing MT, Tracy CR. Do ureteric stent extraction strings affect stent-related quality of life or complications after ureteroscopy for urolithiasis: a prospective randomised control trial. BJU Int. 2014 Apr;113(4):605-9. doi: 10.1111/bju.12541. PMID 24765679
- [Background] Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. BMJ. 1992 Jul 18;305(6846):160-4. doi: 10.1136/bmj.305.6846.160. PMID 1285753
- [Background] Staios D, Andrews HO, Shaik T, Buchholz NN. Quality of life after percutaneous nephrolithotomy for caliceal diverticulum and secluded lower-pole renal stones. J Endourol. 2007 May;21(5):515-9. doi: 10.1089/end.2006.0432. PMID 17523905
- [Background] Joshi HB, Newns N, Stainthorpe A, MacDonagh RP, Keeley FX Jr, Timoney AG. Ureteral stent symptom questionnaire: development and validation of a multidimensional quality of life measure. J Urol. 2003 Mar;169(3):1060-4. doi: 10.1097/01.ju.0000049198.53424.1d. PMID 12576846